CLINICAL TRIAL: NCT01271764
Title: The Association of G9a Protein and Outcome of Patients With Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 099095-E
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Outcome of Endometrial Cancer

ARMS (1):
- endometrial cancer (No Intervention)
  Interventions: Other: no drug

INTERVENTIONS:
Other: no drug — The role of G9a protein in patients with endometrial cancer

SUMMARY:
Tumor invasion and metastasis are the major causes of cancer-related death. Some studies have found that histone methyltransferases, such as EZH2, specifically affect metastasis in breast, gastric and prostate cancer. The functional roles of other members of the HMT family such as G9a in cancer remain obscure. Therefore, the investigators will investigate whether G9a have a role in recurrence/metastasis of endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* all cases with endometrial cancer underwent staging operation

Exclusion Criteria:

* nil

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The role of G9a protein in endometrial cancer | overall survial, disease-free survival
  We will correlate the G9a protein and outcome of endometrial cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan